CLINICAL TRIAL: NCT03573362
Title: Prospective Trial Comparing the Diagnostic Yield of Two Different Needle Sizes Used in EBUS-TBNA for Sarcoidosis and Lymphoma
Brief Title: Effect of Needle Size in Diagnostic Yield of EBUS-TBNA in Sarcoidosis and Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2017-6844
Record Dates: First submitted 2018-05-15; First posted 2018-06-29 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Sarcoidosis; Lymphoma; Adenopathy Hilar
Keywords: sarcoidosis; ebus; endobronchial ultrasound
MeSH Terms: conditions — Sarcoidosis; Lymphoma | interventions — Needles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vizishot Flexneedle 19G (Experimental): Mediastinal and hilar lymph node sampling using the Vizishot Flexneedle19G EBUS-TBNA needle
  Interventions: Device: ViziShot FLEX 19G needle
- Vizishot 22G (Active Comparator): Mediastinal and hilar lymph node sampling using a standard Vizishot 22G EBUS-TBNA needle
  Interventions: Device: Vizishot 22G needle (standard)

INTERVENTIONS:
Device: ViziShot FLEX 19G needle — EBUS-TBNA using the ViziShot FLEX 19G needle
  Arms: Vizishot Flexneedle 19G
Device: Vizishot 22G needle (standard) — EBUS-TBNA using the Vizishot 22G needle (standard)
  Arms: Vizishot 22G

SUMMARY:
The guided FNA by endobronchial ultrasound ( Endobronchial Ultrasound guided transbronchial Needle Aspiration or EBUS-TBNA) is a minimally invasive technique with an established role in the staging of lung cancer 1, and in the evaluation of intrathoracic lymph node metastases from extrathoracic primary cancer2 . There is also a role in cases of isolated hilar and mediastinal lymph nodes in which the differential diagnosis includes mostly sarcoidosis, lymphoma and tuberculosis. 3

Various studies have evaluated more recently the diagnostic yield of EBUS-TBNA specifically for sarcoidosis 4 and thoracic lymphoma 5-6. Although there is emerging data supporting the usefulness of EBUS-TBNA in the investigation of these two pathologies, the efficacy results vary according to the target populations and certain parameters. Moreover, although a large randomized study demonstrated e superiority of EBUS-TBNA over conventional bronchoscopic sampling methods [ bronchoalveolar lavage (BAL) and trans-bronchial biopsies (TBB ] for the diagnosis of sarcoidosis , 7 the results suggest that there is still room for optimizing the performance of EBUS-TBNA [b] . In the field of lymphoma, obtaining large enough specimens for adequate subtyping also remains a concern. 8

In order to improve the performance of EBUS -TBNA , new needles have been developed with the aim to provide biopsies for histological evaluation rather than purely cytological. The ViziShot FLEX © (Olympus) 19 gauge needle (19 gauge or 19G) is a large needle, which can provide both tissue and needle aspiration , and has the advantage of being more flexible.

For this study, the investigators want to compare the diagnostic yield of EBUS-TBNA using needle ViziShot FLEX 19G (1.11 mm) with that of the standard 22G needle ( NA-201SX; Olympus) , in the investigation of hilar or mediastinal lymphadenopathy suspected to be sarcoidosis or lymphoma.

ELIGIBILITY:
Inclusion criteria

* Patient t referred for specimens by EBUS -TBNA with clinical and radiological suspicion of sarcoidosis or lymphoma , with pathological lymph node on imaging (small diameter ≥ 1.0 cm CT-scan or hyper metabolism with PET scan) in para-tracheal stations, sub-carinal and / or hilar (stations 2, 4, 7, 10, 11 and 12), right and / or left.
* Lymph nodes with a small diameter of at least 0.5 cm in CT-scan or PET / CT scan performed in the previous 4-6 weeks.
* Patient investigated in the setting of either an initial diagnosis or a suspicion of lymphoma recurrence (post-treatment).
* Patient able to consent to the procedure and to authorize us by written proxy, included in the consent form for the study, to obtain a copy of the subsequent results or radiological (PET, CT-scan, chest X-ray) or histopathological (linked with age sampled of intrathoracic lymph nodes).
* Patient deemed fit to tolerate the procedure.

Exclusion criteria

* Patient unable to give consent.
* Female patient during pregnancy
* Patient aged under 18.
* Patient with significant coagulopathy ( INR > 1.5 ; platelet count<50 000 / mm 3 ).
* Patient anticoagulated (oral or parenteral) and whose anticoagulation can not be suspended for the procedure.
* Obvious involvement of organ (s) with the possibility of confirming granulomas or suspicious cells of lymphoma by means of a procedure considered less invasive (.. e g, lymph node biopsy of cervical, supraclavicular or inguinal nodes; skin biopsy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of EBUS-TBNA | 12 months after enrollment of the last patient.
  The diagnostic yield of EBUS TBNA with 19G and 22G needle in patients with a final diagnosis of sarcoidosis will be assessed for any difference between the two, using McNemar test on paired proportions.

SECONDARY OUTCOMES:
Ease of use. | 1 week after enrollment of last patient.
  Evaluate the ease of use of both types of needles. Using a visual analog scale (from 0 most difficult to 10 very easy to use), ease of use of each needle will be assessed and compared for each lymph node.
Specimen quality | 1 week after enrollment of last patient
  Samples will be considered adequate if the cytologic assessment shows lymphocytes and or definite if the specimen shows epithelioid cell granulomas or collection of epithelioid cells with a giant cell (or asteroid body or Schaumann body). The samples will be classified as: diagnostic, adequate but non-diagnostic, non-diagnostic and not adequate, no specimen
Complications | 1 month after enrollment of last patient
  Complications encountered with both needle sizes will be compared if there is any difference in the rate of complications, specifically pneumothorax, endobronchial bleeding, post-bronchoscopy bleeding, pneumonia, respiratory infection, hospitalization required because of the procedure, respiratory failure, death.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Vandemoortele, MD, MSc, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided